CLINICAL TRIAL: NCT02434835
Title: Study of Absorption, Metabolism and Excretion Following a Single Oral Dose of [14C]KWA-0711 to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KWA1101
Record Dates: First submitted 2015-04-21; First posted 2015-05-05 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Male Subject

ARMS (1):
- [14C]KWA-0711 (Experimental)
  Interventions: Drug: [14C]KWA-0711

INTERVENTIONS:
Drug: [14C]KWA-0711

SUMMARY:
The purpose of this study is to evaluate the absorption, metabolism and excretion following a single oral dose of [14C]KWA-0711 to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are male, caucasian, and between 35 and 55 years of age, inclusive.
* Subjects who have a body mass index (BMI) between 18.5 and 30.0 kg/m2, inclusive.
* Subjects who have a body weight between 50 and 100 kg, inclusive.
* Subjects must have regular bowel movements.

Exclusion Criteria:

* Subjects who have an abnormality in heart rate, blood pressure , temperature or 12-lead ECG.
* Subjects who are still participating in a clinical study or who have participated in a clinical study involving administration of an investigational drug in the 3 months prior to dose administration.
* Subjects who have had a clinically significant illness within 4 weeks of dose administration as determined by the Investigator.
* Subjects who have any clinically significant abnormal laboratory safety findings.
* Subjects who have had an X ray or who have participated in any clinical trial involving a radiolabelled investigational product or have been exposed to radiolabelled substances within 12 months prior to dose administration.

Ages: 35 Years to 55 Years | Sex: Male
Age Groups: Adult
Dates: Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of total radioactivity, unchanged drug substance and its major metabolites | 240 hours
Maximum observed plasma concentration (Cmax) of total radioactivity, unchanged drug substance and its major metabolites | 240 hours
Cumulative radioactivity recovery in urine and feces | 240 hours
Profiles of metabolites in plasma, urine and faeces | 240 hours

SECONDARY OUTCOMES:
Number of adverse events | 240 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds, United Kingdom